CLINICAL TRIAL: NCT04921865
Title: Observational Case Series on the Clinical Performance of the DePuy Synthes Variable Angle Clavicle Plate and Clavicle Hook Plate 2.7 Systems
Brief Title: Case Series on the Clinical Performance of VA Clavicle and Clavicle Hook Plate 2.7 Systems
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: VA Clavicle
Record Dates: First submitted 2021-05-28; First posted 2021-06-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Clavicle; Acromioclavicular Joint; Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with the DPS VA-LCP® Clavicle Plate 2.7 System or Hook Plate 2.7 System: Any patient undergoing surgical treatment for the fixation of clavicle bone fragments and acromioclavicular joint dislocations using the DPS VA-LCP® Clavicle Plate 2.7 System or DPS VA-LCP® Clavicle Clavicle Hook Plate 2.7 .
  Interventions: Device: DPS VA-LCP® Clavicle Plate 2.7 System; DPS VA-LCP® Clavicle Hook Plate 2.7 System

INTERVENTIONS:
Device: DPS VA-LCP® Clavicle Plate 2.7 System; DPS VA-LCP® Clavicle Hook Plate 2.7 System — The DPS VA-LCP® Clavicle Plate 2.7 System is indicated for the fixation of clavicle bone fragments. The system consists of three plate types: lateral, shaft, and medial, each available in different sizes and materials (titanium alloy and stainless steel). Each plate is available in left and right.
  The DPS VA-LCP® Clavicle Clavicle Hook Plate 2.7 System is indicated or the fixation of lateral clavicle fractures and AC joint dislocations. The Clavicle Hook Plate system consists of three plate types: long, short and button plates.

SUMMARY:
The purpose of this study is to gather early and mid- to long-term evidence to confirm the clinical performance, safety and use of the Clavicle Plate and Clavicle Hook Plate System.

A minimum of 76 patients with clavicle fractures or dislocations of the AC joint surgically treated with any plate from the DPS VA-LCP Clavicle System will be enrolled in this observational post-market clinical investigation.

Outcomes will be collected until up to 2 years after surgery.

DETAILED DESCRIPTION:
Common problems with existing clavicular plates are poor plate 'fit,' unbalance fixation, plate prominence, associated soft tissue irritation, subacromial pain, plate and/or fixation failure (due to unbalanced fixation) and high reoperation rate (for plate removal) [1-3]. The newly developed DePuy Synthes (DPS) variable angle locking compression plate (VA-LCP®) Clavicle 2.7 System was designed to address these problems. The system consists of lateral, shaft and medial plates and hook plates of different sizes to cover a wide variation in clavicular morphology and diverse fracture, fracture-dislocation and dislocation indications.

The objective is to describe the short and long-term clinical performance and safety of both systems, as well as the functional outcomes of this patient population.

Outcomes will be collected at baseline, 2 weeks, 6 weeks, 3 months, 6 months 1, and 2 years after surgery. In addition, the surgeons' experience and utility of the devices will be surveyed. For the short term evaluation, an interim analysis will be done as soon as 30 patients in each group have completed 6 months of follow-up (FU). The final evaluation of long-term outcomes will be done after 2 years of FU.

All treatments and follow-up visits are according to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Unilateral clavicel injury and primary surgical treatment within 21 days from injury with a DPS VA-LCP® Clavicle Plate according to manufacturer's instruction use:

  * VA-LCP® Clavicle Plates 2.7: Fixation of clavicle bone fragments
  * VA-LCP® Clavicle Hook Plates 2.7: Fixation of lateral clavicle fractures and dislocations of the acromioclavicular joint
  * VA-LCP Clavicle Button Hook Plates 2.7: Fixation of acromioclavicular joint dislocations
* Expected ability to attend postoperative FU visits
* Patient informed and consent obtained according to the IRB/EC defined and approved procedures

Exclusion Criteria:

* Stable clavicle fractures
* Systemic infection or infection localized to the site of the proposed implantation
* Concomitant nerve or vessel injury
* Polytrauma (Injury Severity Score ≥ 16)
* BMI ≥40
* Uncontrolled severe systemic disease or terminal illness
* Intraoperative decision to use other implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients treated with the DPS VA-LCP® Clavicle Plate 2.7 System or the DPS VA-LCP® Clavicle Hook Plate 2.7 System for clavicular fracture or dislocations of the acromioclavicular joint
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety aspects | Patients treated with clavicle plate: From baseline up to 24 months after surgery; Patients treated with clavicle hook plate: From baseline until device removal (approximately 3months) and up to 12 months after device removal
  Adverse events (AE) related or possibly related to the investigational device (ADE) or the procedure
Clinical performance | Through study completion, an average of 1 year
  The outcome measures for clinical performance are a subcategory of safety-related parameters (e.g. incidence of complaints related to plate prominence or discomfort, fracture union rate, rate of stable AC joint healing)
Utility in terms of surgeons' experience | Assessed immediately after the surgery
  Surgeons satisfaction with the use and handling of the devices is evaluated in a questionnaire using 5-point Likert scale questions. These include:
  * Surgical time (skin to skin) required for fracture reduction and fixation
    * Much less time than with other implants
    * Slightly less time than with other implants
    * No difference with other implants
    * More time than with other implants
    * Much more time than with other implants
  * Surgeon's impression of the fitting of the device
    * Implant fitted well, no contouring required
    * Implant fitted well, minimal contouring required
    * Implant fitted well laterally but required contouring medially
    * Implant fitted well medially but required contouring laterally
    * Implant required contouring medially and laterally
Surgical time | Assessed immediately after surgeries
  Surgical time in minutes
Fluoroscopy time | Assessed immediately after surgeries
  Fluoroscopy time in minutes
The Disabilities of the Arm Shoulder and Hand short form (QuickDASH) | Patients treated with clavicle plate: From baseline up to 24 months after surgery; Patients treated with clavicle hook plate: From baseline until device removal (approximately 3months) and up to 12 months after device removal
  The Disabilities of the Arm Shoulder and Hand short form (QuickDASH) questionnaire was designed as an occupational health and disability questionnaire. It includes 30 questions that have to be rated from 1 ("no difficulty") to 5 ("unable") where lower values indicate less disability and higher values indicate more disability.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Patients treated with clavicle plate: From baseline up to 24 months after device implantation surgery; Patients treated with clavicle hook plate: From baseline until device removal surgery (approximately 3months) and up to 12 months after device removal
  The PROMIS Physical Function Upper Extremity Short Form 7a v2.0 (2018) consists of 7 questions aimed to evaluate activities that require use of the upper extremity including shoulder, arm, and hand activities. Questions can be rated from 1 "without any difficulties" to 5 "unable to do" where lower values indicate less disability and higher values indicate more disability.

OTHER OUTCOMES:
Patient characteristics | Baseline
  Demographics
Patient characteristics | Baseline
  Height in centimeters
Patient characteristics | Baseline
  Weight in kilograms
Patient characteristics | Baseline
  Body Mass Index (BMI) in kg/m^2
Comorbidities | Baseline
  Concomitant diseases will be assessed using the Charlson Comorbidity Index (CCI). This score assesses the comorbidity level by considering both the number and severity of pre-defined comorbid conditions. It provides a weighted score of a patient's comorbidities which can be used to predict mortality risk. The minimum possible score is 0 (no comorbidities) and maximum 29. The higher the score, the more likely the predicted outcome will result in mortality.
Injury details | Baseline
  Date of injury. Only the year of birth will be assessed.
Injury details | Baseline
  Side injured (i.e. left/right)
Fracture classification | Baseline
  - Clavicle fracture will be recorded using two classifications: AO/OTA Classification and Robinson Classification
  - AC joint dislocation: Rockwood classification
Surgical details | Intraoperative
  Date of surgery
Surgical time | Intraoperative
  Surgical time (i.e. defined as skin-to-skin time) in minutes
Plate details | Intraoperative
  Clavicle Plate System
  * Type of plate and size
    * Lateral
      * CS1
      * CS2
      * CS3
    * Shaft
      * CS1
      * CS2
      * CS3
      * XL
    * Medial
  * Material
    * Stainless steel
    * Titanium alloy
  Clavicle Hook System
  * Type of plate and hook depth
    * Long
      * 9 mm
      * 12 mm
      * 15 mm
    * Short
      * 9 mm
      * 12 mm
      * 15 mm
    * Button
      * 9 mm
      * 12 mm
      * 15 mm
  * Material
    * Stainless steel
    * Titanium alloy
Screw details | Intraoperative
  Screw details will be documented per fragment side (medial and lateral) as:
  * Number of screws
  * Diameter
  * Type
    * variable angle locking
    * metaphyseal
    * cortex
Adjunctive fixations | Intraoperative
  * Osseo cerclage suture
  * Direct ligament suture
  * Internal brace
  * Ligament augmentation for primary repair
  * Suture anchors
  * Muscular reattachment
  * Other
Patient reported outcomes | Patients treated with clavicle plate: From baseline up to 24 months after surgery; Patients treated with clavicle hook plate: From baseline until device removal (approximately 3months) and up to 12 months after device removal
  Pain Numeric Rating Scale (NRS). Local pain will be assessed with the Numerical Rating Scale (NRS). The scale range goes from 0 (no pain) to 10 (worst imaginable pain). A higher value correlates with greater pain.
Radiographical outcomes - Screw density and distribution | Patients treated with clavicle plate: Intraoperative, 2 weeks; Patients treated with clavicle hook plate: Intraoperative, 2 weeks
  Will be assessed in intraoperative or the first postoperative image by analyzing the screw placement with regards to the fracture line, their distribution and type of screws used
Radiographical outcomes - Osteolysis | Patients treated with clavicle hook plate: Intraoperative until device removal (approximately 3months)
  Defined as the presence of a lucent line in the acromion around the tip and body hook of the clavicle hook plate. It will be documented as:
  * Not assessable
  * Partial: any lucency zone around the hook
  * Tip: lucency limited to the tip of the hook
  * Complete: lucency around all zones of the hook
Radiographical outcomes - Bone union | Patients treated with clavicle plate: From baseline up to 24 months after surgery; Patients treated with clavicle hook plate: From baseline until device removal (approximately 3months) and up to 12 months after device removal
  Bone union is defined as the presence of bridging callus in three of four cortices on orthogonal views
Radiographical outcomes - Quality of reduction | Patients treated with clavicle plate: Immediately after surgery; Patients treated with clavicle hook plate: Immediately after surgery
  In cases of fixation failure, quality of reduction will be assessed in the immediate postoperative radiographs and documented as:
  * Accurate reduction of simple fracture
  * Accurate alignment of complex fracture
  * Inaccurate reduction of simple fracture
  * Inaccurate alignment of complex fracture
Radiographical outcomes - Acromioclavicular and coracoclavicular | Patients treated with clavicle plate: From baseline up to 24 months after surgery; Patients treated with clavicle hook plate: From baseline until device removal (approximately 3months) and up to 12 months after device removal
  Acromioclavicular and coracoclavicular distances (in mm) will be assessed using AC joint anteroposterior and Alexander views (if available). The AC distance is the distance between the most medial point on the acromion visible on an anteroposterior view of the AC joint and a point on a line drawn perpendicular to the plane of the dorsal aspect of the lateral or fifth of the clavicle.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lambert, Principal Investigator — University College London Hospital
Locations (7):
- United States (3):
  - Corewell Health, Grand Rapids, Michigan
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
- Klinik Ottakring, Vienna, Austria
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Münster, Münster
- Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] Jaeger M, Sussiek J, Beeres F, Carroll E, Conlan T, Cunningham D, Arnhold R, Lambert S. Observational case series on the clinical performance of the Variable Angle Clavicle Plate and Clavicle Hook Plate 2.7 systems: a study protocol. Front Surg. 2026 Jan 8;12:1694295. doi: 10.3389/fsurg.2025.1694295. eCollection 2025. PMID 41583835